CLINICAL TRIAL: NCT01730274
Title: Cerebellar Tumors of Childhood - Impact on Cognition and Functional Connectivity
Brief Title: Cerebellum - Cognitive Outcome and Functional Connectivity
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christian Dorfer, Dr.med.univ., Medical University of Vienna
Other Study IDs: cerebellum 1.1; KLI 252 (Other Grant/Funding Number: Austrian Science Fund)
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Childhood Cerebellar Tumor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients: children operated on a cerebellar tumor
- healthy subjects: healthy volunteers

SUMMARY:
Aim: To investigate the effect of cerebellar tumor surgery on the resting state functional connectivity level in higher order cognition networks known to interact with the cerebellum. Furthermore, to correlate the connectivity level of these networks with the neuropsychological performance and functional outcome of the patients.

The investigator's hypothesis is that the functional connectivity of various cognition networks in the cerebrum as assessed by resting-state functional magnetic resonance imaging can be impaired after cerebellar tumor surgery and can be correlated with the neuropsychological performance. The effect of surgery on the cognition networks and the neuropsychological performance is dependent on the tumor location within the cerebellum. Such a correlation seems feasible as functional connectivity analysis could be correlated with the neuropsychological impairment in various neuropsychiatric disorders. Furthermore, investigators were able to depict the maturation of the functional connectivity networks in parallel to the neurocognitive development in childhood

ELIGIBILITY:
Inclusion Criteria:

* • Male or female patients aged > 15 yrs

  * Age at surgery between 1 yrs - 12 yrs
  * Compliance (the patients have to be able to lay motionless in a 3 Tesla MR scanner and to cooperate with the examiner during the examination)
  * Signed informed consent from the patient and/or the parents

Exclusion Criteria:

* • Patients with Neurofibromatosis 1

  * Severe visual or auditory impairment
  * Cerebrospinal fluid shunt device
  * Prior radiotherapy or chemotherapy
  * Contraindications to MRI

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: young adolescent operated on a cerebellar tumor as a child
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
neuropsychological assessment | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Dorfer, MD, Principal Investigator — MUV, Department of Neurosurgery
Locations (1):
- MUV, Department of Neurosurgery, Vienna, Austria